CLINICAL TRIAL: NCT06193954
Title: Evaluation of a Vibrational Guidewire System to Facilitate Crossing Coronary Artery Chronic Total Occlusions in Patients With Chronic Angina Refractory to Maximally Tolerated Guideline Directed Medical Therapy
Brief Title: VasoStar Vibrational Guidewire System to Facilitate Crossing Coronary Artery Chronic Total Occlusions
Acronym: VST100
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VasoStar, LLC (Industry)
Collaborators: Summa Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VST100
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Chronic Total Occlusion of Coronary Artery; Chronic Angina

STUDY DESIGN:
Intervention Model Description: Participants may be enrolled in the trial if an attempt to cross the target lesion with a standard wire fails.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- VasoStar guidewire system (Experimental): The VasoStar guidewire system will be used to cross vascular occlusion lesions.
  Interventions: Device: VasoStar guidewire system

INTERVENTIONS:
Device: VasoStar guidewire system — The VasoStar Vibrational Guidewire System vibrates longitudinally at the distal segment of a wire with an electromagnetic source.

SUMMARY:
The goal of this project is to provide an improvement in wire performance to expedite crossing difficult lesions in the coronary vasculature.

DETAILED DESCRIPTION:
This Early Feasibility Study (EFS) is proposed to evaluate the initial safety and efficacy of the VasoStar guidewire system to cross complex coronary vascular lesions in non-tortuous arterial segments which are resistant to crossing with a traditional interventional guidewire.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, over 18 years of age, presenting with at least one ischemia inducing lesion in a native coronary artery that is refractory to standard guidewire crossing. Chronic total occlusion (CTO) is defined as 100% coronary blockage for over a 3-month duration documented either by prior catheterization or by clinical evaluation
* Suitable candidate for non-emergent, coronary angioplasty
* Documented de-novo or restenotic coronary chronic total occlusion defined as a lesion with TIMI 0 flow for at least 90 days refractory to conventional guidewire crossing
* Left ventricle ejection fraction > 20% within the last 12 months.
* For antegrade chronic total occlusion procedures, activated clotting time (ACT) should be > 300 sec
* Chronic total occlusion in a non-tortuous arterial segment
* Voluntarily sign a Patient Informed Consent Form specific to the study.
* Physically and mentally willing to comply with all study requirements.

Exclusion Criteria:

* Successful target lesion crossing with a conventional wire system prior to enrollment
* Prisoners.
* Pregnancy
* Patient has an active implantable.
* Extensive dissection created by refractory guidewire
* Severe ongoing congestive heart failure (New York Heart Association Class IV symptoms)
* Active infection
* Uncontrolled Hypertension (Systolic blood pressure > 180 mm) at the time of the procedure
* History of severe reaction to contrast media
* Recent myocardial infarction (within 2 weeks)
* In-stent target lesion
* Severe cerebrovascular disease including history of prior stroke or transient ischemic attack within 1 month at the time of the procedure
* Saphenous vein graft (SVG) chronic total occlusion or an in-stent chronic total occlusion
* Short life expectancy due to other illnesses such as cancer or pulmonary, hepatic or renal disease
* Participation in another investigational protocol at the time of the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with successful crossing of the target lesion with the VasoStar guidewire system | 1 day
Incidence of Treatment-Emergent Serious Adverse Events | 30 days
  Number of device- or procedure- related serious adverse events

SECONDARY OUTCOMES:
Improved 6-minute walk distance at 6 months following the VasoStar successful procedure | 6 months
Improved 6-minute walk distance at 12 months following the VasoStar successful procedure | 12 months
Improved score on the Seattle Angina Questionnaire at the 6-month visit compared to the score at baseline | 6 months
Improved score on the Seattle Angina Questionnaire at the 12-month visit compared to the score at baseline | 12 months
Reduced number of hospitalizations for cardiac symptoms within 1 year following the VasoStar procedure, compared to the reported number of hospitalizations following standard CTO procedures. | 1 year
Reduced number of emergency room visits for cardiac symptoms within 1 year following the VasoStar procedure, compared to the reported number of hospitalizations following standard CTO procedures. | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Summa Health, Akron, Ohio

IPD SHARING:
Plan to Share IPD: No